CLINICAL TRIAL: NCT02136888
Title: A Single-center, Double-blind, Randomized, Placebo- and Positive-controlled, Parallel-group, Multiple-dose, Up-titration Study of the Electrocardiographic Effects of Ponesimod in Healthy Male and Female Subjects
Brief Title: Study of the Electrocardiographic Effects of Ponesimod in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AC-058-110
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Ponesimod; Safety
MeSH Terms: interventions — ponesimod; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Ponesimod will be administered orally, once daily for 22 days starting on Day 2, and will comprise the following multiple-dose up-titration: 3 days of 10 mg (Days 2 to 4), 3 days of 20 mg (Days 5 to 7), 5 days of 40 mg (Days 8 to 12), 3 days of 60 mg (Days 13 to 15), 3 days of 80 mg (Days 16 to 18), and 5 days of 100 mg (19 to 23).
  Placebo matched for ponesimod will be given on Day -1. Placebo tablets matched for moxifloxacin will be administered on Days 1 and 24.
  Interventions: Drug: Ponesimod Placebo; Drug: Moxifloxacin Placebo; Drug: Ponesimod 10 mg; Drug: Ponesimod 20 mg; Drug: Ponesimod 40 mg; Drug: Ponesimod 60 mg; Drug: Ponesimod 80 mg; Drug: Ponesimod 100 mg
- Group B (Experimental): Placebo matched for ponesimod will be administered orally, once daily on Day -1 and on Day 2 through Day 23. In half of Group B subjects, 400 mg moxifloxacin will be administered orally on Day 1 and a matching placebo tablet on Day 24. In the other half of Group B subjects, a matching placebo tablet will be administered on Day 1 and 400 mg moxifloxacin on Day 24.
  Interventions: Drug: Ponesimod Placebo; Drug: Moxifloxacin Placebo; Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: Ponesimod Placebo
Drug: Moxifloxacin Placebo
Drug: Ponesimod 10 mg
  Other Names: ACT-128800
  Arms: Group A
Drug: Ponesimod 20 mg
  Other Names: ACT-128800
  Arms: Group A
Drug: Ponesimod 40 mg
  Other Names: ACT-128800
  Arms: Group A
Drug: Ponesimod 60 mg
  Other Names: ACT-128800
  Arms: Group A
Drug: Ponesimod 80 mg
  Other Names: ACT-128800
  Arms: Group A
Drug: Ponesimod 100 mg
  Other Names: ACT-128800
  Arms: Group A
Drug: Moxifloxacin 400 mg
  Arms: Group B

SUMMARY:
The aim of this study is to demonstrate that therapeutic and supratherapeutic plasma exposures to ponesimod do not have an effect on cardiac repolarization exceeding the threshold of regulatory concern as measured by the QTc (interval from beginning of the Q wave until end of the T wave corrected for heart rate) interval duration after administration of multiple oral doses of 40 mg and 100 mg to healthy male and female subjects.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, double-blind, randomized, placebo and positive-controlled, double-dummy, parallel group, multiple-dose, up-titration study of the electrocardiographic effects of ponesimod in healthy male and female subjects with a nested cross-over comparison between moxifloxacin and placebo.

Subjects will be randomly assigned to Group A (ponesimod treatment group) or Group B (placebo treatment group) in a 1:1 ratio. Subjects in Group B will be further randomized in a 1:1 ratio to one of the following sequences: 400 mg moxifloxacin followed by moxifloxacin-matching placebo or moxifloxacin matching placebo followed by 400 mg moxifloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Body mass index between 18.0 and 30.0 kg/m^2 (inclusive) at screening.
* Healthy on the basis of medical history and the assessments performed at screening.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to the first drug administration.
* Systolic blood pressure between 90 and 150 mmHg and diastolic blood pressure between 50 and 90 mmHg.
* 12-lead electrocardiogram (ECG) and 24-hour Holter ECG, without clinically relevant abnormalities at screening.
* Hematology and clinical chemistry test results not deviating from the normal range to a clinically relevant extent at screening.
* Negative results from urine drug screen at screening.
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Pregnant or lactating women.
* Known hypersensitivity to moxifloxacin or to any excipients of the drug formulations.
* Veins unsuitable for intravenous puncture on either arm.
* Treatment with another investigational drug within 3 months prior to screening.
* Excessive caffeine consumption, defined as ≥ 800 mg per day at screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study drugs.
* Smoking within 3 months prior to screening.
* Any immunosuppressive treatment within 6 weeks before study drug administration.
* Previous treatment with any prescribed or over-the-counter medications within 2 weeks prior to screening or five half-lives of the drug, whichever is longer.
* Donation of blood, plasma or platelets within 3 months prior to screening or donations made on more than two occasions within the 12 months preceding the first dose administration.
* Lymphopenia (< 1,000 cells/μL^9).
* Viral, systemic, fungal, bacterial or protozoal infection within 4 weeks before the first study drug administration.
* History or clinical evidence suggestive of active or latent tuberculosis at screening.
* Positive hepatitis B surface antigen or hepatitis C antibody tests at screening.
* Positive results from human immunodeficiency virus serology at screening.
* FEV1 or FVC < 80% of the predicted value, or FEV1/FVC ratio < 0.7 at screening.
* History of asthma or chronic obstructive pulmonary disease.
* History of atrioventricular block on ECG.
* Any cardiac condition or illness (including ECG abnormalities based on standard 12-lead ECG or on 24-hour Holter ECG at screening) with a potential to increase the cardiac risk of the subject or that may affect QTc interval analysis.
* QTc interval > 450 milliseconds or > 470 milliseconds for male or female subjects, respectively (using the ECG machine heart rate correction method) at screening.
* Heart rate < 50 beats per minute (bpm) at screening or Day -1 pre-dose on 12-lead ECG.
* Subjects with personal or family history of long QT syndrome or hypokalemia.
* History of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* History or presence of macular edema.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Legal incapacity or limited legal capacity at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted, placebo-corrected effect on QTc interval (time interval from beginning of the Q wave until end of the T wave (ΔΔQTc interval)) on Day 12 (after 5 days of 40 mg ponesimod) | 12 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of ΔΔQTc interval will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 12.
Baseline-adjusted, placebo-corrected effect on QTc interval (time interval from beginning of the Q wave until end of the T wave (ΔΔQTc interval)) on Day 23 (after 5 days of 100 mg ponesimod) | 23 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of ΔΔQTc interval will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 23.

SECONDARY OUTCOMES:
Baseline-adjusted, placebo-corrected effect on QT beat-to-beat interval (QTbtb interval) on Day 12 (after 5 days of 40 mg ponesimod) | 12 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of QTbtb interval will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 12.
Baseline-adjusted, placebo-corrected effect on QT beat-to-beat interval (QTbtb interval) on Day 23 (after 5 days of 100 mg ponesimod) | 23 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of QTbtb interval will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 23.
Baseline-adjusted, placebo-corrected effect on heart rate on Day 12 (after 5 days of 40 mg ponesimod) | 12 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of heart rate will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 12.
Baseline-adjusted, placebo-corrected effect on heart rate on Day 23 (after 5 days of 100 mg ponesimod) | 23 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of heart rate will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 23.
Baseline-adjusted, placebo-corrected effect on the R-to-R interval (interval from the peak of one QRS complex to the peak of the next (RR interval)) on Day 12 (after 5 days of 40 mg ponesimod) | 12 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of RR interval will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 12.
Baseline-adjusted, placebo-corrected effect on the R-to-R interval (interval from the peak of one QRS complex to the peak of the next (RR interval)) on Day 23 (after 5 days of 100 mg ponesimod) | 23 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of RR interval will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 23.
Baseline-adjusted, placebo-corrected effect on the PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) on Day 12 (after 5 days of 40 mg ponesimod) | 12 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of PR interval will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 12.
Baseline-adjusted, placebo-corrected effect on the PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) on Day 23 (after 5 days of 100 mg ponesimod) | 23 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of PR interval will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 23.
Baseline-adjusted, placebo-corrected effect on QRS duration (time interval from the beginning of the Q wave to the end of the S wave) on Day 12 (after 5 days of 40 mg ponesimod) | 12 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of QRS duration will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 12.
Baseline-adjusted, placebo-corrected effect on QRS duration (time interval from the beginning of the Q wave to the end of the S wave) on Day 23 (after 5 days of 100 mg ponesimod) | 23 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of QRS duration will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 23.
Frequency of T-wave morphology changes on Day 12 (after 5 days of 40 mg ponesimod) | 12 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of T-wave morphology changes will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 12.
Frequency of T-wave morphology changes on Day 23 (after 5 days of 100 mg ponesimod) | 23 Days
  Replicate electrocardiograms (ECGs) (at least 3 and up to 10) for the determination of T-wave morphology changes will be extracted from the continuous digital 12-lead ECG recording within 20 minutes prior to dosing and then at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours (total of 13 time points) post-dose on Days -1, 1, and 23.
Change in systolic blood pressure from baseline up to end of study | 31 Days
  Blood pressure will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements should be recorded from the subject in the supine position after having rested for a 5-minute period.
Change in diastolic blood pressure from baseline up to end of study | 31 Days
  Blood pressure will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements should be recorded from the subject in the supine position after having rested for a 5-minute period.
Change in heart rate from baseline up to end of study | 31 Days
  Heart rate will be measured using an automatic oscillometric device, always on the dominant arm (i.e., dominant arm right = writing with right hand). Measurements should be recorded from the subject in the supine position after having rested for a 5-minute period.
Change in QTc interval according to Bazett's correction (QTcB interval) from baseline up to end of study | 31 Days
  QTcB interval will be determined from standard 12-lead ECG recordings. The QTcB interval is the QT interval corrected for heart rate with Bazett's formula (QTcB = QT/RR^0.5 where RR is 60/heart rate)
Change in QTc interval according to Fridericia's correction (QTcF interval) from baseline up to end of study | 31 Days
  QTcF interval will be determined from standard 12-lead ECG recordings. The QTcF interval is the QT interval corrected for heart rate with Fridericia's formula (QTcB = QT/RR^0.5 where RR is 60/heart rate)
Change in forced expiratory volume in 1 second (FEV1) from baseline to end of study | 31 Days
  FEV1 will be measured according to the American Thoracic Society/European Respiratory Society guidelines. Three good test breaths will be measured; the highest FEV1 value will be recorded. The spirometry device must be calibrated and the assessor trained.
Change in forced vital capacity (FVC) from baseline to end of study | 31 Days
  FVC will be measured according to the American Thoracic Society/European Respiratory Society guidelines. Three good test breaths will be measured; the highest FVC value will be recorded. The spirometry device must be calibrated and the assessor trained.
Incidence of treatment emergent pulmonary function test decreases of >30% from baseline up to end of study | 31 Days
  Pulmonary function tests will be performed according to the American Thoracic Society/European Respiratory Society guidelines. Three good test breaths will be measured; the highest values will be recorded. The spirometry device must be calibrated and the assessor trained.
Area under the plasma concentration-time curve of ponesimod from time zero over the dosing interval (τ) (AUCτ) after 5 days of dosing with 40 mg ponesimod | 12 Days
  Plasma concentrations of ponesimod will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 12 (after 5 days of dosing with 40 mg ponesimod). AUCτ will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification (LOQ).
Maximum plasma concentration (Cmax) of ponesimod after 5 days of dosing with 40 mg ponesimod | 12 Days
  Plasma concentrations of ponesimod will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 12 (after 5 days of dosing with 40 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain Cmax.
Time to maximum plasma concentration (tmax) of ponesimod after 5 days of dosing with 40 mg ponesimod | 12 Days
  Plasma concentrations of ponesimod will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 12 (after 5 days of dosing with 40 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain tmax.
Trough plasma concentration of ponesimod on Days 5, 8, 16, and 19 (Ctrough) | 19 Days
  Plasma concentrations of ponesimod will be measured on Days 5, 8, 16, and 19 immediately before administration of the study drug.The measured individual plasma concentrations will be used to directly obtain Ctrough.
Area under the plasma concentration-time curve of the ponesimod metabolite ACT-204426 from time zero over the dosing interval (τ) (AUCτ) after 5 days of dosing with 40 mg ponesimod | 12 Days
  Plasma concentrations of ACT-204426 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 12 (after 5 days of dosing with 40 mg ponesimod). AUCτ will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification (LOQ).
Maximum plasma concentration (Cmax) of the ponesimod metabolite ACT-204426 after 5 days of dosing with 40 mg ponesimod | 12 Days
  Plasma concentrations of ACT-204426 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 12 (after 5 days of dosing with 40 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain Cmax.
Time to maximum plasma concentration (tmax) of the ponesimod metabolite ACT-204426 after 5 days of dosing with 40 mg ponesimod | 12 Days
  Plasma concentrations of ACT-204426 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 12 (after 5 days of dosing with 40 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain tmax.
Area under the plasma concentration-time curve of the ponesimod metabolite ACT-338375 from time zero over the dosing interval (τ) (AUCτ) after 5 days of dosing with 40 mg ponesimod | 12 Days
  Plasma concentrations of ACT-338375 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 12 (after 5 days of dosing with 40 mg ponesimod). AUCτ will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification (LOQ).
Maximum plasma concentration (Cmax) of the ponesimod metabolite ACT-338375 after 5 days of dosing with 40 mg ponesimod | 12 Days
  Plasma concentrations of ACT-338375 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 12 (after 5 days of dosing with 40 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain Cmax.
Time to maximum plasma concentration (tmax) of the ponesimod metabolite ACT-338375 after 5 days of dosing with 40 mg ponesimod | 12 Days
  Plasma concentrations of ACT-338375 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 12 (after 5 days of dosing with 40 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain tmax.
Area under the plasma concentration-time curve of ponesimod from time zero over the dosing interval (τ) (AUCτ) after 5 days of dosing with 100 mg ponesimod | 23 Days
  Plasma concentrations of ponesimod will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 23 (after 5 days of dosing with 100 mg ponesimod). AUCτ will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification (LOQ).
Maximum plasma concentration (Cmax) of ponesimod after 5 days of dosing with 100 mg ponesimod | 23 Days
  Plasma concentrations of ponesimod will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 23 (after 5 days of dosing with 100 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain Cmax.
Time to maximum plasma concentration (tmax) of ponesimod after 5 days of dosing with 100 mg ponesimod | 23 Days
  Plasma concentrations of ponesimod will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 23 (after 5 days of dosing with 100 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain tmax.
Area under the plasma concentration-time curve of the ponesimod metabolite ACT-204426 from time zero over the dosing interval (τ) (AUCτ) after 5 days of dosing with 100 mg ponesimod | 23 Days
  Plasma concentrations of ACT-204426 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 23 (after 5 days of dosing with 100 mg ponesimod). AUCτ will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification (LOQ).
Maximum plasma concentration (Cmax) of the ponesimod metabolite ACT-204426 after 5 days of dosing with 100 mg ponesimod | 23 Days
  Plasma concentrations of ACT-204426 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 23 (after 5 days of dosing with 100 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain Cmax.
Time to maximum plasma concentration (tmax) of the ponesimod metabolite ACT-204426 after 5 days of dosing with 100 mg ponesimod | 23 Days
  Plasma concentrations of ACT-204426 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 23 (after 5 days of dosing with 100 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain tmax.
Area under the plasma concentration-time curve of the ponesimod metabolite ACT-338375 from time zero over the dosing interval (τ) (AUCτ) after 5 days of dosing with 100 mg ponesimod | 23 Days
  Plasma concentrations of ACT-338375 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 23 (after 5 days of dosing with 100 mg ponesimod). AUCτ will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification (LOQ).
Maximum plasma concentration (Cmax) of the ponesimod metabolite ACT-338375 after 5 days of dosing with 100 mg ponesimod | 23 Days
  Plasma concentrations of ACT-338375 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 23 (after 5 days of dosing with 100 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain Cmax.
Time to maximum plasma concentration (tmax) of the ponesimod metabolite ACT-338375 after 5 days of dosing with 100 mg ponesimod | 23 Days
  Plasma concentrations of ACT-338375 will be measured at pre-dose and at 1, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 11, and 12 hours post-dose on Day 23 (after 5 days of dosing with 100 mg ponesimod). The measured individual plasma concentrations will be used to directly obtain tmax.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Brossard, PhD, Study Director — Actelion
Locations (1):
- Covance Clinical Research Unit (CRU), Evansville, Indiana, United States

REFERENCES:
- [Derived] Hoch M, Darpo B, Brossard P, Zhou M, Stoltz R, Dingemanse J. Effect of ponesimod, a selective S1P1 receptor modulator, on the QT interval in healthy individuals. Basic Clin Pharmacol Toxicol. 2015 May;116(5):429-37. doi: 10.1111/bcpt.12336. Epub 2014 Nov 8. PMID 25287214